CLINICAL TRIAL: NCT01785147
Title: Randomized Placebo Controlled Trial Assessing the Efficacy and Safety of BP1.4979 in Smoking Cessation
Brief Title: Efficacy and Safety of BP1.4979 in Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P12-01 / BP1.4979; 2012-002731-28 (EudraCT Number)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Tobacco Addiction
Keywords: Tobacco addition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- BP1.4979 3mg (Experimental): BP1.4979 3mg during 3 months
  Interventions: Drug: BP1.4979
- BP1.4979 10mg (Experimental): BP1.4979 10mg during 3 months
  Interventions: Drug: BP1.4979
- BP1.4979 15mg (Experimental): BP1.4979 15mg during 3 months
  Interventions: Drug: BP1.4979
- Placebo (Placebo Comparator): Placebo during 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP1.4979 — BP1.4979 at 3mg, 10mg, 15mg or placebo during 3 months.
  Arms: BP1.4979 10mg; BP1.4979 15mg; BP1.4979 3mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
Clinical study which aim is to assess in heavy smokers willing to quit smoking the efficacy and the safety profile of BP1.4979 for smoking cessation on the total abstinence measured by subject diary and confirmed by exhaled CO (abstinent < 10 ppm).

DETAILED DESCRIPTION:
BP1.4979 is a novel compound with promising efficacy on smoker which have been assessed on phase I studies.

This is a multicenter,randomized, double blind, placebo controlled, phase IIb trial with parallel group to assess safety and efficacy of BP1.4979 in smoker.

ELIGIBILITY:
Main inclusion Criteria:

* a smoking history of at least 10 years
* subject smoking at least 15 cigarettes per day at the time being and for at least 30 days before selection.
* having already made at least 2 attempts to stop
* with no period of abstinence > 3 months in the previous year
* FTND ≥ 7

Main exclusion Criteria:

* any significant psychiatric illness or mood disorder, assessed by the BDI
* HAD scale (A + D ≥ 19, the day of the selection and inclusion)
* AUDIT ≥ 8
* subject smoking cigars or pipes exclusively
* subject taking any antismoking medication and/ or Nicotine Replacement Therapy (NRT) in the previous month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
4-week prolonged abstinence from smoking cigarettes | 4 weeks
  The primary measure of efficacy will be 4-week prolonged abstinence from smoking cigarettes at the end of 12-week double-blind treatment phase (i.e. from V3 to V4).
  The continuous abstinence measured by subject diary and verified by exhaled CO (abstinent < 10 ppm) will define response to the treatment.

SECONDARY OUTCOMES:
7-day tobacco Point Prevalence Abstinence (PPA) | 7 days
  7-day tobacco Point Prevalence Abstinence (PPA) will be assessed at each visit by analysis of cigarettes consumption using self-report diaries and measurement of exhaled CO
Number of adverse events | 26 weeks
  Assessment of safety thanks to the number and clinical evaluation of the adverse events.
Vital signs measures | 26 weeks
  Vital signs (measurement of heart rate, blood pressure, and body weight) will be assessed at each study visit, thanks to physical examinations (V0 and V4), ECG and laboratory tests (blood chemistry, haematology, urinanalysis tests, prolactin dosage) at screening (V0), after 4-week treatment (V2) and at V4.

CONTACTS AND LOCATIONS:
Overall Officials: Henri-Jean AUBIN, MD, Ph.D, Principal Investigator — Hôpital Paul Brousse
Locations (1):
- Hôpital Paul Brousse, Villejuif, Île-de-France Region, France